CLINICAL TRIAL: NCT01396070
Title: Exploratory Pilot Study of Brentuximab Vedotin (SGN-35) in Patients With Mycosis Fungoides and Sézary Syndrome With Variable CD30 Expression Level
Brief Title: Brentuximab Vedotin (SGN-35) in Patients With Mycosis Fungoides With Variable CD30 Expression Level
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Youn Kim (Other)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor-Investigator, Youn Kim, The Joanne and Peter Haas, Jr, Professor for Cutaneous Lymphoma Research, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-21324; LYMNHL0089 (Other: OnCore); SU-06212011-7946 (Other: Stanford University)
Record Dates: First submitted 2011-07-14; First posted 2011-07-18 (Estimated); Results first posted 2017-04-05 (Actual); Last update posted 2017-04-05 (Actual); Status verified 2017-02

CONDITIONS: Non-Hodgkin Lymphoma (NHL); Cutaneous Lymphoma; Cutaneous T-cell Lymphoma (CTCL); Mycosis Fungoides; Sezary Syndrome
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Brentuximab vedotin (Experimental): Novel antibody-drug conjugate, 1.8 mg/kg intravenously every 3 weeks
  Interventions: Drug: Brentuximab vedotin

INTERVENTIONS:
Drug: Brentuximab vedotin — 1.8 mg/kg by IV every 3 weeks for a maximum of 16 doses (8 cycles).
  Brentuximab vedotin is an antibody conjugate, consisting of the chimeric IgG1 anti-CD30 antibody cAC10; the microtubule disrupting agent monomethyl auristatin E (MMAE); a protease-cleavable linker that covalently attaches MMAE to cAC10.
  Other Names: Adcetris; SGN-35

SUMMARY:
The purpose of this study is to learn the effects of brentuximab vedotin (SGN-35), an investigational medication, on patients with cutaneous T cell lymphoma (CTCL), specifically mycosis fungoides (MF) and Sezary syndrome (SS). Despite a wide range of therapeutic options, the treatments are associated with short response duration, thus this condition is largely incurable. This investigational drug may offer less toxicity than standard treatments and have better tumor specific targeting.

DETAILED DESCRIPTION:
This phase 2 exploratory study will evaluate the clinical response of brentuximab vedotin in MF and SS, where tumor cells express variable levels of CD30 target molecule.

The primary objective is to explore the biologic activity of brentuximab vedotin in patients with MF and SS, the most common types of cutaneous T-cell lymphoma (CTCL), where expression of CD30 is variable. Brentuximab vedotin has significant biologic activity in Hodgkin's disease (HD) where only a small numbers of CD30 positive tumor cells are present, as well as in lymphomas with large numbers of CD30-expressing tumor cells such as systemic anaplastic large cell lymphoma (sALCL). The subject grouping by CD30 expression levels (low, intermediate, high) is for accrual purposes only, to ensure that a wide range of CD30 expression is studied.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven MF/SS, stage IB-IVB, and failed one standard systemic therapy. Skin biopsy must be within 3 months of beginning study medication
* At least the following wash-out from prior treatments:

  * ≥ 3 weeks for local radiation therapy, systemic cytotoxic anticancer therapy, treatment with other anti-cancer investigational agents (including monoclonal antibody)
  * > 3 weeks for retinoids, interferons, vorinostat, romidepsin, denileukin diftitox and phototherapy
  * > 2 wks for topical therapy (including topical steroid, retinoid, nitrogen mustard, or imiquimod)
* At least 18 years of age
* ECOG performance status of ≤ 2
* Must be able to commit to study schedule
* Absolute neutrophil count (ANC) ≥ 1000/uL
* Platelets ≥ 50,000/uL
* Bilirubin ≤ 2X upper limit of normal (ULN) (EXCEPTION: Gilbert's disease ≤ 3X ULN)
* Serum creatinine ≤ 2X ULN
* Alanine aminotransferase (ALT) ≤ 3X ULN
* Aspartate aminotransferase (AST) ≤ 3X ULN
* Negative serum beta-HCG pregnancy test result within 7 days of first treatment, if a woman of childbearing potential
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Mycosis fungoides (MF) with limited disease (stage IA) or central nervous system (CNS) disease
* Systemic or topical concomitant corticosteroid use for treatment of skin disease (EXCEPTION: Oral prednisone allowed at ≤ 10 mg/day)
* Known Grade 3 or higher (per NCI CTCAE v4.0 criteria) active systemic or cutaneous viral, bacterial, or fungal infection
* Known to be Hepatitis B or Hepatitis C antibody positive
* HIV-positive with have a measurable viral load while on antiretroviral medication
* Known hypersensitivity to recombinant proteins or any excipient contained in the drug formulation.
* History of other malignancies during the past 3 years (EXCEPTIONS: non-melanoma skin cancer; curatively treated localized prostate cancer; curatively treated localized breast cancer; resected thyroid cancer; cervical intraepithelial neoplasia; or cervical carcinoma in situ on biopsy).
* Pregnant
* Breastfeeding
* Congestive heart failure, Class III or IV, by New York Heart Association (NYHA) criteria.
* Any serious underlying medical condition that would impair subject's ability to receive or tolerate the planned treatment.
* Dementia or altered mental status that would preclude subject's understanding and rendering of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-05; Primary Completion 2015-04 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Youn H Kim, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim YH, Tavallaee M, Sundram U, Salva KA, Wood GS, Li S, Rozati S, Nagpal S, Krathen M, Reddy S, Hoppe RT, Nguyen-Lin A, Weng WK, Armstrong R, Pulitzer M, Advani RH, Horwitz SM. Phase II Investigator-Initiated Study of Brentuximab Vedotin in Mycosis Fungoides and Sezary Syndrome With Variable CD30 Expression Level: A Multi-Institution Collaborative Project. J Clin Oncol. 2015 Nov 10;33(32):3750-8. doi: 10.1200/JCO.2014.60.3969. Epub 2015 Jul 20. PMID 26195720

RESULTS

PARTICIPANT FLOW:
Groups:
- Brentuximab Vedotin: Brentuximab vedotin 1.8 mg/kg intravenously (IV) once every 3 weeks (1 cycle)
Period: Overall Study
Arm/Group | Brentuximab Vedotin
Started | 36
Completed | 17
Not Completed | 19
Not completed — Withdrawal by Subject | 2
Not completed — Death | 2
Not completed — Adverse Event | 8
Not completed — Physician Decision | 3
Not completed — Lack of Efficacy | 4

BASELINE CHARACTERISTICS:
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 33
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 25
  More than one race | 0
  Unknown or Not Reported | 4
CD30 grouping at screening [Number; unit: participants] — Level of CD30 expression was defined at the % CD30 positivity in the total lymphocytic infiltrate, stratified as 0 to < 10% ; 10% to 50%; or over 50%.
  participants
    < 10% CD30 positivity | 17
    10% to 50% CD30 positivity | 15
    > 50% CD30 positivity | 4
Clinical Stage [Count of Participants; unit: Participants] — MF/SS staging is based on a tumor-node-metastasis-blood (TNMB) classification system. The most important prognostic factors include overall clinical stage, T-classification, and extracutaneous disease.
  Early stage includes MF IA, IB, and IIA. Advanced stage includes MF IIB and higher, including MF/SS IVA.
  Participants
    Stage IB | 6
    Stage IIB | 16
    Stage IV/SS (includes IVA, IVA/SS and III) | 14

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Overall response rate of brentuximab vedotin in this study population.
Time Frame: 2 years
Population: The percentage was calculated by adding Complete response (CR) + Partial Response (PR) = Overall rate. 3 subjects were not evaluable.
Measure: Number; unit: percentage
Groups:
- Overall Response Rate (%): Overall Response Rate of all patients
Arm/Group | Overall Response Rate (%)
Number analyzed (Participants) | 33
percentage
  Everyone evaluable (ORR) | 70
  Tissue CD30 Expression Group A: number analyzed (Participants) | 16
  Tissue CD30 Expression Group A | 56
  Tissue CD30 Expression Group B: number analyzed (Participants) | 14
  Tissue CD30 Expression Group B | 79
  Tissue CD30 Expression Group C: number analyzed (Participants) | 3
  Tissue CD30 Expression Group C | 100
  Stage IB: number analyzed (Participants) | 5
  Stage IB | 83
  Stage IIB: number analyzed (Participants) | 20
  Stage IIB | 94
  Stage IV/SS: number analyzed (Participants) | 8
  Stage IV/SS | 63
  Females: number analyzed (Participants) | 11
  Females | 30
  Males: number analyzed (Participants) | 22
  Males | 69

2. Secondary Outcome: Overall Stable Disease Rate
Description: Overall Stable Disease Rate (SD) in this study population.
  3 subjects were not evaluable.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 33
Participants | 5

3. Secondary Outcome: Overall Partial Response Rate
Description: Overall Partial Response Rate (PR) in this study population.
  3 subjects were not evaluable.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 33
Participants | 21

4. Secondary Outcome: Overall Non-Evaluable Response
Description: Overall Non-Evaluable Response of full patient population
  3 subjects were not evaluable.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Brentuximab Vedotin
Number analyzed (Participants) | 33
Participants | 4

ADVERSE EVENTS:
Time Frame: 4 weeks
Groups:
- All Participants: All reported AE's on trial
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 23/36
Other Adverse Events (participants affected / at risk) | 32/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=36)
Sepsis (Infections and infestations) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Blood disorder (Blood and lymphatic system disorders) | 2 (5)
Skin Infection (Infections and infestations) | 2 (2)
Confusion (Psychiatric disorders) | 1 (1)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 (2)
Hypercalcemia (Blood and lymphatic system disorders) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (4)
Pneumonia (Reproductive system and breast disorders) | 1 (1)
GVHD (Gastrointestinal disorders) | 1 (1)
White blood cell decreased (Blood and lymphatic system disorders) | 1 (1)
Acute kidney Injury (Gastrointestinal disorders) | 1 (2)
Infection and Pain of skin (Musculoskeletal and connective tissue disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Vomitting (Gastrointestinal disorders) | 1 (1)
Hypomagnesemia (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=36)
Peripheral Neuropathy (Nervous system disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 3 (3)
Skin eruption (Skin and subcutaneous tissue disorders) | 4 (4)
Weight Loss (Social circumstances) | 3 (3)
Aberrant T-cell population (blood) (Blood and lymphatic system disorders) | 2 (2)
Dysphonia (Blood and lymphatic system disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hyponatremia (Blood and lymphatic system disorders) | 2 (2)
Infusion Reaction (General disorders) | 2 (2)
Leukopenia (Investigations) | 2 (2)
Lower extremity edema (General disorders) | 2 (2)
LFTs elevated (Investigations) | 2 (2)
Myalgias (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No